CLINICAL TRIAL: NCT02040610
Title: A Phase II Study of Hypofractionated Image Guided Proton Therapy for Low and Intermediate Risk Prostate Cancer
Brief Title: Hypofractionated Image Guided Proton Therapy for Low andIntermediate Risk Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Provision Center for Proton Therapy (Other)
Collaborators: Center for Biomedical Research, LLC (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO 1401; NCT02198222 (obsolete NCT alias)
Record Dates: First submitted 2014-01-16; First posted 2014-01-20 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Prostate Cancer
Keywords: Low Risk Prostate Cancer; Intermediate Risk Prostate Cancer; Hypofractionated; Image Guided Proton Therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Proton Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low Risk Prostate Cancer (Active Comparator): Hypofractionated Proton Therapy 62 Gy (RBE) in 20 fractions of 3.1 Gy (RBE) over 4 weeks
  Interventions: Radiation: Hypofractionated Proton Therapy
- Intermediate Risk Prostate Cancer (Active Comparator): Hypofractionated Proton Therapy 62 Gy (RBE) in 20 fractions of 3.1 Gy (RBE) over 4 weeks
  Interventions: Radiation: Hypofractionated Proton Therapy

INTERVENTIONS:
Radiation: Hypofractionated Proton Therapy
  Other Names: Proton Therapy

SUMMARY:
This study is being proposed to evaluate the use of moderate hypofractionated proton therapy in low and intermediate risk prostate cancer patients. Quality of life outcomes as well as gastrointestinal and genitourinary early and late toxicities will be analyzed and compared to conventional proton therapy regimens. It is thought that this regimen will produce comparable findings and would result in substantial health care cost savings, as well as, be more convenient for patients.

DETAILED DESCRIPTION:
Patients will receive: 62 Gy (RBE) in 20 fractions of 3.1 Gy (RBE) over 4 weeks

ELIGIBILITY:
Inclusion Criteria:

* Pathological (histologically) proven diagnosis of prostatic adenocarcinoma within 365 days (1 year) prior to study registration.

  * History and physical exam with digital rectal exam of the prostate to establish clinical staging
  * Clinical stage T1-T2c (AJCC 7th edition) within 90 days of registration.
  * Prostate specific antigen (PSA) < 20 ng/mL within 90 days prior to registration.
  * Gleason Score < 7.
  * Eastern Cooperative Oncology Group(ECOG) Performance status 0-1.
  * Clinically negative lymph nodes evaluated by imaging (pelvic +/- abdominal CT or MRI scan).
  * Patients with lymph nodes equivocal or questionable by imaging are eligible without biopsy if the nodes are ≤ 1.5 cm in diameter; any node larger than this on imaging will require negative biopsy for eligibility, unless the node is know to be enlarged from prior scans and considered stable, per discretion of the treating physician.
  * Patients must be 18 years of age or older.
  * Patient must be able to provide study-specific informed consent prior to study entry.
  * Willingness and ability to complete the Expanded Prostate Cancer Index Composite (EPIC) Questionnaire.
  * No evidence of bone metastases (M0) on bone scan within 60 days prior to registration.
  * Bone scan is not required for patients enrolled with a single intermediate risk factor only, but this scan may be obtained at the discretion of the treating physician. Patients with 2 or 3 risk factors will require a negative bone scan for eligibility.
  * Equivocal bone scan findings are allowed if plain film x-rays are negative for metastasis.
  * Patient is able to start proton therapy or neo-adjuvant hormonal therapy, when recommended, within 12 weeks of registration.
  * No prior radiotherapy to the pelvic area.
  * No prior prostate cancer therapy such as: prostatectomy, cryotherapy, chemotherapy or hyperthermia.
  * Platelets ≥ 100,000 cells/mm3, Absolute neutrophil count (ANC) ≥ 1,800 cells/mm3, Hemoglobin ≥ 8.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dl is acceptable.)
  * Obs.: Patients with high risk factors, such as T3, Gleason 8-10 or PSA > 20ng/mL who are not considered candidates for pelvic lymph node radiation treatment are still considered eligible for this study.

Exclusion Criteria:

* • Prior radiotherapy to the pelvic area.

  * Prior prostate cancer therapy such as: prostatectomy, cryotherapy, or hyperthermia.
  * Prior systemic therapy (chemotherapy) for prostate cancer.
  * Evidence of distant metastases.
  * Regional lymph node involvement.
  * Previous or concurrent cytotoxic chemotherapy for prostate cancer.
  * Acquired Immune Deficiency Syndrome (AIDS) based upon current Centers for Disease Control (CDC) definition. Note however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive. Protocol-specific requirements may also exclude immune-compromised patients.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Estimated)
Dates: Start 2014-01; Primary Completion 2019-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Time to biochemical failure | 5 years
  To determine the freedom from biochemical failure survival outcomes (FFBF) and compare to historical FFBF results achieved following standard fractionation proton therapy

SECONDARY OUTCOMES:
Toxicity Assessment | 2 years & 5 years
  To determine the incidence of acute and late Gastrointestinal and Genitourinary toxicity at 2 and 5 years.
Analyze Quality of Life | 2 years & 5 years
  To assess quality of life following proton therapy (QOL EPIC) at 2 and 5 years

OTHER OUTCOMES:
Salvage Androgen Deprivation Therapy | Every 6 months for 5 years
  To determine the need for salvage Androgen Deprivation Therapy for biochemical or other relapse events

CONTACTS AND LOCATIONS:
Overall Officials: J. Ben Wilkinson, M.D., Principal Investigator — Provision Center for Proton Therapy
Locations (2):
- United States (2):
  - Provision Cares Proton Therapy Center Knoxville, Knoxville, Tennessee
  - Provision Cares Proton Therapy Center Nashville, Nashville, Tennessee